CLINICAL TRIAL: NCT03384238
Title: A Phase I/II Study Evaluating the Safety and Pharmacokinetics of Panitumumab-IRDye800 as an Optical Imaging Agent to Detect Pancreas Cancer During Surgical Procedures
Brief Title: Panitumumab-IRDye800 in Patients With Pancreatic Cancer Undergoing Surgery
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eben Rosenthal (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Professor of Otolaryngology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-42237; NCI-2017-01943 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PANC0028 (Other: OnCore); R01CA190306 (NIH)
Record Dates: First submitted 2017-12-19; First posted 2017-12-27 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Optical Imaging; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1a (Experimental): A test/loading dose of 100 mg of unlabeled Panitumumab (fixed dose) will be administered via a 60 minute IV infusion prior to infusion of the Panitumumab IRDye800. Cohort 1a will receive 25 mg of Panitumumab IRDye800 with a 100 mg unlabeled test/loading dose of Panitumumab. The surgical resection will then occur 2 to 5 days after infusion. Intraoperative imaging will be performed using the intraoperative optical imaging devices
  Interventions: Procedure: Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800
- Cohort 1b (Experimental): Cohort 1b will receive 50 mg of Panitumumab IRDye800 with a 100 mg unlabeled test/loading dose of Panitumumab. A test/loading dose of 100 mg of unlabeled Panitumumab (fixed dose) will be administered via a 60 minute IV infusion prior to infusion of the Panitumumab IRDye800. The surgical resection will then occur 2 to 5 days after infusion. Intraoperative imaging will be performed using the intraoperative optical imaging devices
  Interventions: Procedure: Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800
- Cohort 1c (Experimental): Cohort 1c will receive 75 mg of Panitumumab IRDye800 with a 100 mg unlabeled test/loading dose of Panitumumab.A test/loading dose of 100 mg of unlabeled Panitumumab (fixed dose) will be administered via a 60 minute IV infusion prior to infusion of the Panitumumab IRDye800. The surgical resection will then occur 2 to 5 days after infusion. Intraoperative imaging will be performed using the intraoperative optical imaging devices
  Interventions: Procedure: Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800
- Cohort 1d (Experimental): Cohort 1d will receive a 50 mg dose of Panitumumab IRDye800 and no test/loading dose. A test/loading dose of 100 mg of unlabeled Panitumumab (fixed dose) will be administered via a 60 minute IV infusion prior to infusion of the Panitumumab IRDye800. The surgical resection will then occur 2 to 5 days after infusion. Intraoperative imaging will be performed using the intraoperative optical imaging devices
  Interventions: Procedure: Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800
- Cohort 2- Dose Expansion (Experimental): Cohort 2 will receive the optimal dose of Panitumumab-IRDye800 as determined in Cohort 1
  Interventions: Procedure: Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800

INTERVENTIONS:
Procedure: Fluorescence Imaging — Undergo fluorescence imaging
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix
Drug: Panitumumab-IRDye800 — Given IV
  Other Names: Panitumumab IRDye 800; RDye800-Panitumumab Conjugate

SUMMARY:
This phase I/II trial studies the side effects and best dose of panitumumab-IRDye800 and to see how well it works in finding cancer in patients with pancreatic cancer who are undergoing surgery. Panitumumab-IRDye800 is a combination of the antibody drug panitumumab and IRDye800CW, an investigational dye that can be seen using a special camera. Panitumumab-IRDye800 may attach to tumor cells and make them more visible during surgery in patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the optimal dose of panitumumab-IRDye800 in identifying pancreatic cancer compared to surrounding normal tissue in the ex vivo setting as measured by tumor to background ratio.

SECONDARY OBJECTIVES:

I. Determine the safety and tolerability of the panitumumab-IRDye800 as an imaging agent in subjects undergoing resection of pancreatic cancer.

II. Determine whether metastatic lesions, positive lymph node, or residual disease can be detected by near-infrared (NIR) fluorescence imaging with panitumumab-IRDye800 but not by white light.

OUTLINE: This is a phase I, dose-escalation study of panitumumab-IRDye800 followed by a phase II study.

Patients receive a loading dose of panitumumab intravenously (IV) over 60 minutes, and after 15 minutes of observation, patients then receive panitumumab-IRDye800 IV over 60 minutes on day 0. Patients then undergo surgical resection 2-5 days after panitumumab-IRDye800 administration with imaging using the Novadaq SPY/LUNA, Novadaq IR9000 fluorescence imaging system with open field handheld fluorescence imaging camera, and/or pinpoint endoscopic fluorescence imaging camera, and SurgVision Explorer Air multi spectral fluorescence reflectance system.

After completion of study treatment, patients are followed up at 15 and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected or biopsy-confirmed diagnosis of pancreatic adenocarcinoma
* Planned standard of care surgery with curative intent for pancreatic adenocarcinoma
* Life expectancy of more than 12 weeks
* Karnofsky performance status of at least 70% or Eastern Cooperative Oncology Group (ECOG)/Zubrod level =< 1
* Hemoglobin >= 9 gm/dL
* Platelet count >= 100,000/mm^3
* Magnesium > the lower limit of normal per institution normal lab values
* Potassium > the lower limit of normal per institution normal lab values
* Calcium > the lower limit of normal per institution normal lab values
* Thyroid-stimulating hormone (TSH) < 13 micro international units/mL

Exclusion Criteria:

* Received an investigational drug within 30 days prior to first dose of panitumumab-IRDye800
* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); or unstable angina within 6 months prior to enrollment
* History of infusion reactions to panitumumab or other monoclonal antibody therapies
* Pregnant or breastfeeding
* Evidence of corrected QT (QTc) prolongation on pretreatment electrocardiography (ECG) (greater than 440 ms in males or greater than 460 ms in females)
* Lab values that in the opinion of the physician would prevent surgical resection
* Patients receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Tumor to background ratio (TBR) | 1 day
  TBR is defined as fluorescence intensity of tumor tissue compared to that of normal surrounding pancreatic tissue.

SECONDARY OUTCOMES:
Number of Grade 2 or higher AEs determined to be clinically significant and definitely, probably or possibly related to study drug | Up to 30 days
  Safety events will be recorded over the 30 day observation period.
Number of positive lymph nodes per participant, not detected by white light | 1 day
  Determine whether positive lymph nodes can be detected by near-infrared (NIR) fluorescence imaging with Panitumumab-IRDye800 but not by white light.
Number of positive resection margins per participant, not detected by white light | 1 day
  Determine whether residual disease at resection margins can be detected by near-infrared (NIR) fluorescence imaging with Panitumumab-IRDye800 but not by white light.

CONTACTS AND LOCATIONS:
Overall Officials: George Poultsides, Principal Investigator — Stanford University; Eben Rosenthal, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu G, van den Berg NS, Martin BA, Nishio N, Hart ZP, van Keulen S, Fakurnejad S, Chirita SU, Raymundo RC, Yi G, Zhou Q, Fisher GA, Rosenthal EL, Poultsides GA. Tumour-specific fluorescence-guided surgery for pancreatic cancer using panitumumab-IRDye800CW: a phase 1 single-centre, open-label, single-arm, dose-escalation study. Lancet Gastroenterol Hepatol. 2020 Aug;5(8):753-764. doi: 10.1016/S2468-1253(20)30088-1. Epub 2020 May 14. PMID 32416764